CLINICAL TRIAL: NCT02580565
Title: PHEDRE Trial Protocol - Observational Study of the Prevalence of Problematic Use of Equimolar Mixture of Oxygen and Nitrous Oxide (EMONO) and Analgesics in the French Sickle-cell Disease Population
Brief Title: Prevalence of Problematic Use of Equimolar Mixture of Oxygen and Nitrous Oxide and Analgesics in the Sickle-cell Disease
Acronym: PHEDRE
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: University Hospital, Marseille (Other); University Hospital, Clermont-Ferrand (Other); University Hospital, Toulouse (Other); University Hospital, Paris (Other); University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: RC14_0344
Record Dates: First submitted 2015-09-28; First posted 2015-10-20 (Estimated); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Sickle Cell Disease
Keywords: sickle cell disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: telephone interview — Clinical assessment for screening and a phone call for questionnaire administration

SUMMARY:
The use of analgesics can lead to cases of drug abuse and dependence. It can also cause pseudo-addiction in patients suffering from pain. What is the actual situation in patients suffering from severe sickle-cell disease, exposed to acute pain during vaso-occlusive crises? Evaluation of the use of analgesics, on the basis of Diagnostic and Statistical Manual of Mental Disorders criteria for substance abuse and dependence, makes it possible to differentiate the symptoms occurring only in a context of pain, in the aim of managing the pain, and thus describing pseudo-addiction, from symptoms also occurring when there is no pain, and more in favour of true addiction. Currently there is no data available in France on this problem, and no studies have been carried out in children or adolescents with sickle-cell disease. The purpose of the study is to evaluate the prevalence of problematic use of equimolar mixture of oxygen and nitrous oxide and other analgesic drugs in a population of subjects with severe sickle-cell disease in France.

PHEDRE (Pharmacodépendance Et DREpanocytose-drug dependence and sickle-cell disease) is an observational, descriptive and transversal study. Patients under the age of 26 with sickle-cell disease are included in the study by the doctors looking after them in sickle-cell disease centres. The patients are then contacted by a trained researcher for a telephone interview, including an evaluation of the Diagnostic and Statistical Manual of Mental Disorders criteria for abuse and dependence to equimolar mixture of oxygen and nitrous oxide and for each of the analgesic drugs taken by the patient. The data are also completed using the subject's medical record.

This study will make it possible to provide an initial quantitative and qualitative evaluation of problematic use of equimolar mixture of oxygen and nitrous oxide and analgesic drugs in the sickle-cell disease population. The results will be used firstly to provide additional data essential for monitoring the risk of overdose, abuse, dependence and misuse of these products, and to begin awareness-raising and to provide information for health care professionals, in order to significantly improve the management of sickle-cell disease-related pain.

DETAILED DESCRIPTION:
This is a national multicentric observational study

•Clinical assessment

After he includes a patient, the medical practitioner complete a clinical assessment which contains all information about patient's family and personal history, history of the SCD and treatment already received for SCD. The clinical assessment is kept in the Reference Centre or Special Centre for Children and Adults (RSCCA). Therefore, the trained researcher will schedule a visit to the RSCCA to retrieve the clinical assessments of all patients included in this RSCCA and enter the data in the electronic case report form (e-CRF).

* Telephone interview

Telephone interview is carried out with a trained researcher from Nantes CEIP-A. When Nantes CEIP-A receipts the inclusion form and written consent, the trained researcher schedules a telephone interview with the patient. The interview is suited to the child's, adolescent's or young adult's age, maturity and comprehension skills. The following parameters are evaluated during the telephone semi-structured interview for EMONO, and for other analgesic drugs, during pain episodes and outside pain episodes.

ELIGIBILITY:
Inclusion Criteria:

* Subject with confirmed SCD diagnosis, regardless whether it is the homozygous or heterozygous form
* Subject treated for SCD at a RSCCA participating in the study, regardless of the duration of the illness
* Subject under the age of 26
* Written consent from adult subjects and written consent from one of the parents or legal guardians of minors

Exclusion Criteria:

* State-protected adult (under guardianship)
* Subject not having the general aptitude to participate in the study assessment (i.e. not able to respond to the telephone interview): too young, insufficient motor development, major difficulties understanding the French language and/or speech and/or hearing disorders

Ages: 6 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: French sickle-cell disease population who has a problematic use of Equimolar Mixture of Oxygen and Nitrous Oxide (EMONO) and analgesics
Sampling Method: Non-Probability Sample
Enrollment: 1004 (Actual)
Dates: Start 2015-09-25 (Actual); Primary Completion 2016-09-25 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Problematic use is abuse of or dependence on a substance according to the fourth edition of DSM (DSM-IV), and substance use disorder according to the fifth edition (DSM 5). | 24 months after the start of the study
  The primary outcome mesure is evaluation of problematic use of EMONO. The DSM (Diagnostic and Satistical Manual) identifies 11 criteria for problematic use. The presence or absence of each criteria is assessed by phone with the patient. Therefore, the total number of criteria is calculated for each patient and represents the severity of problematic use.

CONTACTS AND LOCATIONS:
Overall Officials: Marie GERARDIN, Doctor, Principal Investigator — Hospital practitioner

REFERENCES:
- [Derived] Gerardin M, Rousselet M, Couec ML, Masseau A; PHEDRE Group; Aquizerate A, Authier N, Deheul S, Roussin A, Micallef J, Djezzar S; French Addictovigilance Network (FAN); Feuillet F, Jolliet P, Grall-Bronnec M, Victorri-Vigneau C. Substance use disorder of equimolar oxygen-nitrous oxide mixture in French sickle-cell patients: results of the PHEDRE study. Orphanet J Rare Dis. 2024 Mar 18;19(1):124. doi: 10.1186/s13023-024-03133-w. PMID 38500184
- [Derived] Gerardin M, Rousselet M, Couec ML, Masseau A, Guerlais M, Authier N, Deheul S, Roussin A, Micallef J, Djezzar S; French Addictovigilance Network (FAN); Feuillet F, Jolliet P, Victorri-Vigneau C. Descriptive analysis of sickle cell patients living in France: The PHEDRE cross-sectional study. PLoS One. 2021 Mar 18;16(3):e0248649. doi: 10.1371/journal.pone.0248649. eCollection 2021. PMID 33735176
- [Derived] Gerardin M, Couec ML, Grall-Bronnec M, Feuillet F, Wainstein L, Rousselet M, Pinot ML, Perrouin F, Bonnot O, Drouineau MH, Jolliet P, Victorri-Vigneau C. PHEDRE trial protocol - observational study of the prevalence of problematic use of Equimolar Mixture of Oxygen and Nitrous Oxide (EMONO) and analgesics in the French sickle-cell disease population. BMC Psychiatry. 2015 Nov 14;15:281. doi: 10.1186/s12888-015-0677-5. PMID 26573686